CLINICAL TRIAL: NCT03481439
Title: Improving Medication Safety: Development and Impact of Multivariate Model-based Strategy to Target High-risk Patients of Postoperative Complication
Brief Title: Development and Impact of Multivariate Model-based Strategy to Target High-risk Patients of Postoperative Complication
Acronym: HiRisP3
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0134
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-03

CONDITIONS: Orthopaedic Surgery; Traumatology
Keywords: Pharmacist; Led medication review; Orthopaedic surgery; Traumatology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary cohort: Primary cohort : Cohort of patient between January and February 2017
  Interventions: Other: Collection of a Pharmaceutical intervention
- Secondary cohort: Secondary cohort : Cohort of patient between February and March 2018
  Interventions: Other: Collection of a Pharmaceutical intervention

INTERVENTIONS:
Other: Collection of a Pharmaceutical intervention — collection of pharmaceutical interventions carried out by the pharmaceutical team in the care uni in Primary and secondary cohort

SUMMARY:
The objective is therefore to create a risk score for ADEs in an orthopedic and traumatological surgery department.

The study is an prospective, observational, cohort trial. A first step will consist of: (i) a collection of PIs carried out in an orthopedic and traumatological surgery department for 1 month, (ii) a score of the clinical impact of Pharmacist Interventions using the Clinical, Econnomic and organisationnal scale by method of consensus and (iii) a statistical analysis. Statistical analysis consists of (i) logistic regression modeling, (ii) performance measurement by discrimination and calibration, and internal validation by resampling. In a second step, external validation using a new sample will be performed.

DETAILED DESCRIPTION:
Pharmaceutical means for clinical pharmacy activities and pharmaceutical analysis are limited. Several methods can be used to increase the efficiency of resources allocated to clinical pharmacy activities. We hypothesize that highlighting patients at risk for iatrogenic drug events (ADEs) by applying a predictive score of ADE could be a way to increase the efficiency of clinician pharmacist interventions.

b. Assumption (s) and objective (s) The use of a predictive score of ADE in hospitalized patients in orthopedic surgery would make it possible to prioritize clinical pharmacy actions according to the resources allocated. The objective is therefore to create a risk score for ADEs in an orthopedic and traumatological surgery department. The secondary objective is to evaluate its superiority over other predictive models such as the age or the Physical Status Score physical status score used by anesthetists.

c. Methodology The study is an prospective, observational, cohort trial. A first step will consist of: (i) a collection of PIs carried out in an orthopedic and traumatological surgery department for 1 month, (ii) a score of the clinical impact of Pharmacist Interventions (NPS) using the Clinical, Econnomic and organisationnal scale by method of consensus and (iii) a statistical analysis. Statistical analysis consists of (i) logistic regression modeling, (ii) performance measurement by discrimination and calibration, and internal validation by resampling. In a second step, external validation using a new sample will be performed.

d. Expected results and prospects The usefulness of clinical pharmacy activities is now demonstrated, however an improvement in their efficiency is needed. The prospects are the integration of the risk score in the dispensing assistance software connected to the computerized patient record as well as extending the score to other types of surgery.

ELIGIBILITY:
Inclusion criteria:

* Subject aged over 18 years
* Subject hospitalized in the department of orthopaedic surgery and traumatology on university hospital of Montpellier.

Exclusion criteria:

* Vulnerable persons according to French law (pregnant women, adults under guardianship, persons deprived of liberty)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient hospitalized in the department of orthopaedic surgery and traumatology on university hospital of Montpellier
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Major clinical impact pharmaceutical intervention | 1 day
  Occurrence of a major clinical impact pharmaceutical intervention according to the CLEO scale

SECONDARY OUTCOMES:
pharmaceutical intervention | 1 day
  Occurrence of a pharmaceutical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pierre RENAUDIN, Pharm D, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
Not determined